CLINICAL TRIAL: NCT01397695
Title: Topical Bevacizumab for the Management of Recurrent Epistaxis in Patients With Hereditary Hemorrhagic Telangiectasia (HHT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090666
Record Dates: First submitted 2011-07-18; First posted 2011-07-19 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Hereditary Hemorrhagic Telangiectasia (HHT)
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bevacizumab (Experimental)
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — The bevacizumab will then be sprayed by the treating physician in the clinic, under direct observation. Spray will be achieved by administering the bevacizumab through a mucosal atomization device. 0.1cc will be sprayed into both nares. Patients will then sit for 5 minutes, the application will be repeated for a total of 40 applications, thereby administering 50mgs into each nostril, a total of 100mgs into each patient. The 5 minute spacing has been arbitrarily chosen as sufficient time for 0.1cc of solution to be absorbed by the nasal mucosa. That will complete the treatment.

SUMMARY:
Terence M. Davidson, MD is conducting a research study to find out more about the topical application of Avastin (proper chemical name is bevacizumab) in the treatment of epistaxis (nose bleeding) in patients with Hereditary Hemorrhagic Telangiectasia (HHT).

DETAILED DESCRIPTION:
Plans are to recruit patients with HHT from the UCSD Nasal Dysfunction Clinic. The HHT world is connected through the HHT Foundation. The Foundation is interested in VEGF inhibitors. They have carefully watched our work at UCSD for a long time and our two papers on Avastin have been circulated around the world. Those who come for our evaluation and are deemed appropriate for Bevacizumab injection will be recruited for this study. Those agreeing to participate will sign a consent form.

The treatment, regardless of participation in the proposed research, is to bring the patients to the operating room where under general anesthesia the nose is suctioned clean of blood clot, crust and secretion. The mucosa is then injected with a local anesthetic with adrenaline to reduce discomfort and to reduce bleeding. The nasal mucosa is treated with a KTP laser in our standard fashion. A 100mg of Avastin delivered in 4cc is then diluted with 4cc of normal saline to a total volume of 8cc. The dilution is made not for any known difference in treatment but rather it normally takes a minimum of 8cc to properly inject the nasal mucosa. The 1% Bevacizumab is then injected submucosally throughout the nasal cavity sparing the mucosa of the cartilage and the septum. The nasal cavity is then sprayed with 2cc of a fibrin sealant (EVICEL) this reduces postoperative bleeding and facilitates healing from the laser therapy. It has nothing to do with the Bevacizumab injection. The patient is then awakened and returned to the recovery room and discharged home. Beginning in approximately one week the patient is instructed to begin their hypertonic pulsatile nasal irrigations. They will follow-up in the clinic at 1 month. The data collection form is attached. Prior to treatment patient completes the HHT epistaxis severity score, blood is drawn for hematocrit, hemoglobin and serum feritin levels. Women of childbearing age all have a urine pregnancy test, required both by anesthesia and for the Bevacizumab study as well. Patients are followed monthly for the first 6 months. At 3 and 6 months the blood tests are repeated. For those living in San Diego they can be performed at UCSD. For those living outside the San Diego area they can be repeated by their primary care physician. For the ensuing 18 months patients are followed monthly either electronically or by telephone. ESS scores are calculated. Laboratory tests are not repeated. Patients are followed-up until such time as they begin re-bleeding and their ESS scores increase either above 2 or by 1 point above their 1 month post-op evaluation. Experience to date with 20 or 30 patients is that bleeding ceases within 1 to 2 weeks. Hence the 1 month score should be their optimum result. Adverse events will be recorded and appropriately reported to the IRB.

A new epistaxis severity score (ESS) has been developed and tested by the HHT Foundation. We have used this for the past several months and found it to be an excellent measure of HHT epistaxis. A copy is attached.

The minimum sample size is 10 patients. Study duration is planned for 24 months and if more patients are recruited they will be included. If fewer patients are recruited the study may be extended. Data will be reported by means and standard deviations. Patients will be compared individually and collectively to their pretreatment data specifically hematocrit, hemoglobin, serum ferritin and epistaxis severity score. All medical information collected at UCSD will be included in their EPIC electronic medical record. All data will be maintained on a de-identified spreadsheet. Patients will be numbered 1-99. A separate database correlating patient number with name and medical record number will be kept separately. Both of these data sheets are maintained on a password protected computer and backed-up on a thumb drive. These are maintained within the University Medical Center and a locked office.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 18
* Both male and non-pregnant females adults capable of making informed consent who have HHT by Curacao criteria and whose nasal bleeding due to HHT is of such a magnitude that it requires medical care
* Additionally, females of childbearing age will be given a pregnancy test as a preliminary measure to ensure that those who become involved are not at risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terence Davidson, M.D., Principal Investigator — UCSD
Locations (1):
- University of California, San Diego Medical Center, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Responsible Party for this record has passed away in 2013. There are no study team members still associated with this study at the institution. There have been no publications, and the study data cannot be located.
Period: Overall Study
Arm/Group | Bevacizumab
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Responsible Party for this record has passed away in 2013. There are no study team members still associated with this study at the institution. There have been no publications, and the study data cannot be located.
Arm/Group | Bevacizumab
Number analyzed (Participants) | 0
Age, Categorical
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Epistaxis in Patients With HHT as Measured by the HHT Foundation Epistaxis Severity Score, Hematocrit, Hemoglobin and Serum Ferritin Levels.
Description: The Responsible Party for this record has passed away in 2013. There are no study team members still associated with this study at the institution. There have been no publications, and the study data cannot be located.
Time Frame: 1-2 years
Population: as for baseline characteristics
Arm/Group | Bevacizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The Responsible Party for this record has passed away in 2013. There are no study team members still associated with this study at the institution. There have been no publications, and the study data cannot be located.
Arm/Group | Bevacizumab
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes